CLINICAL TRIAL: NCT05446298
Title: Phase 2 Randomized Open-label Multicenter Study of Combination of ONC-392 and Pembrolizumab for the Treatment of Patients With Platinum Resistant Ovarian Cancer (PROC)
Brief Title: ONC-392 and Pembrolizumab in Platinum Resistant Ovarian Cancer
Acronym: PRESERVE-004
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESERVE-004; KEYNOTE-E24 and MK3475-E24 (Other: Merck Sharp & Dohme LLC); GOG-3081 (Other: GOG Partners); 20224734 (Other: WCG IRB)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; High Grade Serous Adenocarcinoma of Ovary; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 mg/kg ONC-392 and 200 mg pembrolizumab (Experimental): Arm A: Pembrolizumab 200 mg will be administered by IV infusion over 30 minutes, followed by ONC-392 at 1.0 mg/kg will be administered by IV infusion over 60 minutes, q3w.
  Interventions: Drug: ONC-392; Drug: Pembrolizumab
- 2 mg/kg ONC-392 and 200 mg pembrolizumab (Experimental): Arm B: Pembrolizumab 200 mg will be administered by IV infusion over 30 minutes, followed by ONC-392 at 2.0 mg/kg will be administered by IV infusion over 60 minutes, q3w.
  Interventions: Drug: ONC-392; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ONC-392 — ONC-392 will be given by IV infusion, q3w.
  Other Names: A humanized anti-CTLA4 IgG1 monoclonal antibody made by OncoC4, Inc.
Drug: Pembrolizumab — Pembrolizumab in fixed dose of 200 mg will be given by IV infusion, q3w.
  Other Names: MK3475; Keytruda

SUMMARY:
This is a study to test the safety and efficacy with the combination of a next generation anti-CTLA-4 antibody, ONC-392, and anti-PD-1 antibody, pembrolizumab, in platinum resistant ovarian cancer patients.

DETAILED DESCRIPTION:
The purpose of this Phase 2 study is to compare two doses of ONC-392 in combination with a fixed dose of pembrolizumab in participants with ovarian cancer who are resistant to platinum-based chemotherapy and have disease progression on line of therapy containing bevacizumab. Results from this study will be used to inform the study design, patient population, and dose selection for future studies in advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yrs old female patients who provide written informed consent for the study.
2. Patients must have a confirmed diagnosis of high-grade serous ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
3. Patients must have received prior standard of care of surgical intervention, including hysterectomy and salpingo-oophorectomy.
4. Patients must have platinum-resistant disease:

   1. Patients who have only 1 line of systemic therapy must have completed a minimum of four cycles of platinum-based therapy with CR or PR and then progressed between 3 to 6 months after the last dose of platinum.
   2. Patients who have received 2 or more lines of platinum therapy must have progressed ≤ 6 months (183 days) after the last dose of platinum.

   The time is calculated from the date of last administrated dose of platinum therapy to the date of radiographic imaging with disease progression.
5. Patients must have received 1 or more prior systemic lines of anti-cancer therapy with or without bevacizumab or a PARP inhibitor, and for whom single-agent therapy is appropriate as the next line of treatment:

   1. Adjuvant ± neoadjuvant is considered 1 line of therapy
   2. Maintenance therapy (eg, bevacizumab, PARP inhibitors) will be considered part of the preceding line of therapy (ie, not counted independently)
   3. Therapy changed due to toxicity in the absence of progression will be considered part of the same line (ie, not counted independently)
   4. Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance.
6. At least 1 measurable target lesion according to RECIST 1.1, including the following criteria:

   1. Non-nodal lesion that measures ≥1.0 cm in the longest diameter
   2. Lymph node (LN) lesion that measures as ≥1.5 cm in the short axis
   3. The lesion is suitable for repeat measurement using computed tomography/magnetic resonance imaging (CT/MRI). Lesions that have had external beam radiotherapy (EBRT) or locoregional therapy must show radiographic evidence of subsequent growth.
7. ECOG score 0 or 1.
8. Time from prior therapy:

   1. Systemic anti-cancer therapy (5 half-lives of small molecule drugs or 4 weeks, whichever is shorter)
   2. Focal radiation completed at least 2 weeks prior to first dose of study drug.
   3. Major surgery must be completed at least 4 weeks prior to first dose of study drug. Patients have recovered or stabilized from the adverse effects of the prior surgery.
9. In the opinion of the investigator, the patient must have a life expectancy of at least 12 weeks and is well enough to receive experimental therapy.
10. Adequate organ function as determined by laboratory tests as defined below at screening.

System Laboratory Value Hematological Absolutely neutrophil count (ANC) ≥1500/µL Platelets ≥100,000/µL Hemoglobin1 ≥9.0 g/dL or 5.6 mmol/L Renal Creatinine clearance as calculated per Cockcroft-Gault or MDRD formula > 30 mL/min Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN except for unconjugated hyperbilirubinemia of Gilbert's syndrome.

AST, ATL ≤3 × ULN (≤5 × ULN for participants with liver metastases) Serum Albumin ≥ 2.5 g/dL

Exclusion Criteria:

1. Patients with carcinosarcoma (malignant mixed Mullerian tumor), clear cell carcinoma, endometrioid, low grade serous, clear cell, and mucinous adenocarcinoma, and ovarian cancer not otherwise specified.
2. Patients with primary platinum-refractory disease, defined as disease that did not respond to (CR or PR), or has progressed within 3 months of the last dose of first-line platinum-containing chemotherapy.
3. Patients who are at high risk for disease progression including those who have ascites requiring a paracentesis within 14 days before first treatment.
4. Patients with active symptomatic CNS metastases, unless they have received local therapy (e.g., whole brain radiation therapy [WBRT], surgery or radiosurgery) 21 days before study treatment and have discontinued the use of corticosteroids for this indication for a minimum of 7 days prior to study treatment.
5. Patients who are on chronic systemic steroid therapy for autoimmune conditions or as immunosuppression at doses higher than 10 mg/day prednisone or equivalent within 7 days before first treatment.
6. Active second malignancy with anti-cancer treatments (except for treated in-situ carcinomas [e.g., breast, cervix, bladder], or basal or squamous cell carcinoma of the skin) within the past 24 months. HIV patient with Karposi sarcoma or Castleman disease will be excluded. Patient with renal cell carcinoma will be excluded.
7. Prior history of symptomatic pulmonary embolism or significant cardiovascular impairment within 12 months of the first dose of study drug: such as history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, or cerebrovascular accident (CVA) stroke, or cardiac arrhythmia associated with hemodynamic instability.
8. Active infection requiring systemic IV antibiotics or hospitalization within 14 days prior to administration of study drugs. Regular treatment of urinary tract infection (UTI) and/or topical treatment are allowed.
9. Patients who have not recovered to CTCAE V5.0 Grade 0 or 1 (except chemotherapy related peripheral neuropathy in Grade 2 or less, or endocrinopathy with adequate replacement therapy) from any toxicity and/or complications from major surgery or prior cancer therapeutics before starting therapy. The hemoglobulin criteria must be met without packed RBC transfusion within 14 days of study treatment.
10. Any evidence of current interstitial lung disease (ILD) or pneumonitis, or a prior history of ILD or non-infectious pneumonitis that required steroid treatment.
11. Patients who have active inflammatory bowel disease or intestinal obstruction.
12. Patients who, in the opinion of the Investigator, have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, have mental health issues that might interfere with the patient's participation for the full duration of the study or make study participation, or not in the best interest of the patient. The Investigator should discuss with the Sponsor and/or study leaders.
13. Participating in other clinical trials or receiving other anti-cancer therapy. Patient who has prior anti-PD-1, PD-L1, or CTLA-4 antibody based therapies will be excluded.
14. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Administration of killed vaccines are allowed.
15. Patient who had an allogenic tissue/organ transplant or stem cell transplantation will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  To assess the efficacy of ONC-392 and pembrolizumab combination therapy in objective response rate per RECIST1.1.
Treatment Related Adverse Events (TRAEs) and Immune Related Adverse Events (irAEs) | 24 months
  To assess the safety of ONC-392 and pembrolizumab combination therapy

SECONDARY OUTCOMES:
Duration of Response (DoR) | 24 months
  To assess the efficacy of ONC-392 and pembrolizumab combination therapy measured by duration of response.
Disease Control Rate (DCR) | 24 months
  To assess the efficacy of ONC-392 and pembrolizumab combination therapy measured by DCR.
Best Overall Response (BOR) | 24 months
  To assess the efficacy of ONC-392 and pembrolizumab combination therapy measured by BOR.
Progression Free Survival (PFS) | 24 months
  PFS as assessed by BICR according to RECIST 1.1 and iRECIST.
Overall Survival (OS) | 24 months
  OS as assessed from randomization to the time the subject expired.
Pharmacokinetics and exposure-response analysis | 24 months
  Drug concentration measurement in relation to safety and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Monk, MD, Principal Investigator — GOG Partners; Joyce Barlin, MD, Principal Investigator — GOG Partners
Locations (21):
- United States (21):
  - Cancer Treatment Centers of America, Phoenix. 403, Goodyear, Arizona
  - Honor Health, USOR, 406, Phoenix, Arizona
  - Nuvance Health System, 401, Danbury, Connecticut
  - Baptist MD Anderson Cancer Center, 404, Jacksonville, Florida
  - Sudarshan Sharma, MD. LTD. 414, Hinsdale, Illinois
  - Cancer Treatment Centers of America, Chicago. 410, Zion, Illinois
  - Northwest Cancer Centers - Dyer, IN - USOR, 422, Dyer, Indiana
  - Baptist Health Lexington, 407, Lexington, Kentucky
  - Norton Cancer Institute - St. Matthews, 416, Louisville, Kentucky
  - Willis-Knighton Physician Network / Gynecologic Oncology Associates, 409, Shreveport, Louisiana
  - Minnesota Oncology Hematology, P. A. - USOR, 421, Maplewood, Minnesota
  - Center of Hope, 413, Reno, Nevada
  - The Valley Hosptial, Inc. 411, Ridgewood, New Jersey
  - Women's Cancer Care Associates, LLC. 405, Albany, New York
  - The Ohio State University James Cancer Center, 412, Columbus, Ohio
  - Oncology Associates of Oregon, P. C. - USOR. 419, Eugene, Oregon
  - Texas Oncology, P. A. - Austin, USOR. 417, Austin, Texas
  - Texas Oncology, P.A., Fort Worth - USOR. 420, Fort Worth, Texas
  - Texas Oncology, P. A. Woodlands - USOR, 418, The Woodlands, Texas
  - Texas Oncology - Northeast Texas - USOR, 423, Tyler, Texas
  - Medical College of Wisconsin, 408, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Du X, Liu M, Tang F, Zhang P, Ai C, Fields JK, Sundberg EJ, Latinovic OS, Devenport M, Zheng P, Liu Y. Hijacking antibody-induced CTLA-4 lysosomal degradation for safer and more effective cancer immunotherapy. Cell Res. 2019 Aug;29(8):609-627. doi: 10.1038/s41422-019-0184-1. Epub 2019 Jul 2. PMID 31267017
- [Background] Du X, Liu M, Su J, Zhang P, Tang F, Ye P, Devenport M, Wang X, Zhang Y, Liu Y, Zheng P. Uncoupling therapeutic from immunotherapy-related adverse effects for safer and effective anti-CTLA-4 antibodies in CTLA4 humanized mice. Cell Res. 2018 Apr;28(4):433-447. doi: 10.1038/s41422-018-0012-z. Epub 2018 Feb 20. PMID 29463898
- [Background] Barlin JN, Lim PC, Thomes Pepin J, Hopp EE, Cloven NG, Lee C, Eshed HD, Black D, Cottrill HM, Hand L, O'Malley DM, Chuang LT, Willmott L, Chisamore M, Shpyro S, Durbin J, Zheng P, Liu Y, Monk BJ. LBA32 A randomized, phase II, dose optimization of gotistobart, a pH-sensitive anti-CTLA-4, in combination with standard dose pembrolizumab in platinum-resistant recurrent ovarian cancer: Safety, efficacy and dose optimization (PRESERVE-004/GOG-3081). Annals of Oncology, 2024. 35: p. S1224-S1225. doi: 10.1016/j.annonc.2024.08.2271
- [Background] Barlin JN, Lim PC, Thomes Pepin J, Hopp EE, Cloven NG, Eshed HD, Black D, Cottrill HM, Hand L, O'Malley DM, Chuang LT, Chisamore M, Durbin J, Zheng P, Liu Y, Shpyro S, Monk BJ.LB010/#1590 A phase 2 randomized dose optimization trial of gotistobart, a PH-sensitive anti-CTLA-4, in combination with pembrolizumab in platinum-resistant ovarian cancer (PROC, preserve-004/GOG-3081; NCT05446298). International Journal of Gynecological Cancer, 2024. 34: p. A6-A8. doi: 10.1136/ijgc-2024-IGCS.7